CLINICAL TRIAL: NCT01180543
Title: Phase II- Acne Treatment With Active Patches Which Contains Azelaic Acid, Citric Acid,Salicylic Acid and 2% Ascorbic Acid
Brief Title: Acne Treatment With Active Oplon's Patches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oplon-Pure Science Ltd. (Industry)
Responsible Party: Avner Shemer M.D., Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP002
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator: Oplon Active Patch (Active Comparator)
  Interventions: Device: Oplon Active Patch
- Placebo Comparator: Placebo patch (Placebo Comparator)
  Interventions: Device: Placebo Patch

INTERVENTIONS:
Device: Oplon Active Patch — Patches are placed over acne lesion overnight. Treatment is a single treatment.
  Arms: Active Comparator: Oplon Active Patch
Device: Placebo Patch — same as active patch
  Arms: Placebo Comparator: Placebo patch

SUMMARY:
The purpose of this study was to demonstrate the effect of short treatment with active OPLON patches on Acne.

DETAILED DESCRIPTION:
Patients with Acne Vulgaris were treated overnight with active patches. Effect is observed at the end of the treatment and 24 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Acne Vulgaris
* Over 18 years
* Signing informed consent

Exclusion Criteria:

* Active treatment of acne
* Change in hormonal therapy
* Antibiotic treatment in a week prior to the experiment
* Sensitive skin
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Severity Score of lesion | Severity Score of lesion [Time Frame: 24 hours following patch removal]
  Lesions were ranked by investigator according to severity whereas:
  0-clear, 1-mild, 2-moderate, 3-sever

SECONDARY OUTCOMES:
Severity Score of lesion | Severity Score of lesion [Time Frame: 12 hours with the patch]
  Lesions were ranked by investigator according to severity whereas:
  0-clear, 1-mild, 2-moderate, 3-sever

CONTACTS AND LOCATIONS:
Overall Officials: Avner Shemer, M.D., Principal Investigator — Laniado Medical Center
Locations (1):
- Dermatology Clinic, Netanya, Israel